CLINICAL TRIAL: NCT00370513
Title: A Phase I, Open-Label, Dose-Escalation, Multi-Center Study or Pazopanib (GW786034) in Adult Patients With Hepatocellular Cancer
Brief Title: A Phase I Study of Pazopanib in Adult Patients With Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG107200
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: pazopanib; liver cancer; hepatocellular cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — pazopanib

ARMS (1):
- Pazopanib Arm (Experimental): Different doses of oral pazopanib once daily for the duration of the study starting on Day 1 of Treatment Period 1. Treatment continues until disease progression or withdrawl from study.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — Pazopanib is a potent, multi-target receptor tyrosine kinase inhibitor of VEGFR.

SUMMARY:
Liver cancer is a good target for anti-angiogenic treatments such as pazopanib. The effect of pazopanib in patients with liver cancer are unknown. This study is designed to evaluate the safety, tolerability and best dose of pazopanib to be given to patient with liver cancer.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of advanced liver cancer adequate bone marrow, liver and kidney function
* Any local therapy for tumor must have been completed at least 4 weeks prior to enrolling in study

Exclusion criteria:

* Pregnant or breastfeeding
* Any serious or unstable medical or psychiatric conditions
* History of metastases to central nervous system
* History of ulcer, inflammatory bowel disease or disease of the gut
* History of HIV, or uncontrolled infection
* Have had a cardiac condition or stoke during the past 6 months
* High blood pressure
* Have had a blood clot during the past 6 months
* History of bleeding blood vessels

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-12-06 (Actual); Primary Completion 2009-04-08 (Actual); Study Completion 2009-04-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and changes in vital signs and laboratory values. A dose regimen where no more than 1 out of 6 subjects experience a dose-limiting toxicity (DLT) will define the maximum tolerated dose (MTD). | throughout the study

SECONDARY OUTCOMES:
Various pharmacokinetic parametersAlpha-fetoprotein (AFP) measurements and scans | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, San Francisco, California, United States
- GSK Investigational Site, Hong Kong, Hong Kong
- GSK Investigational Site, Taipei, Taiwan

REFERENCES:
- [Background] Yau T, Chen PJ, Chan P, Curtis CM, Murphy PS, Suttle AB, Gauvin J, Hodge JP, Dar MM, Poon RT. Phase I dose-finding study of pazopanib in hepatocellular carcinoma: evaluation of early efficacy, pharmacokinetics, and pharmacodynamics. Clin Cancer Res. 2011 Nov 1;17(21):6914-23. doi: 10.1158/1078-0432.CCR-11-0793. Epub 2011 Aug 10. PMID 21831954
- See also: Results for study VEG107200 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG107200?search=study&search_terms=107200#rs